CLINICAL TRIAL: NCT00720018
Title: A Phase I, Single Center, Open Label, Single-Dose, Five-Period Study to Compare the Pharmacokinetics of NP101 (Sumatriptan Iontophoretic Transdermal Patch) in Healthy Volunteers
Brief Title: Phase I Open Label Single-Dose Study to Compare the Pharmacokinetics of NP101 Healthy Volunteers
Acronym: NP101-006
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NuPathe Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PROT-15-NP101-006
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Period 1 (Experimental): NP101 Patch
  Interventions: Drug: NP101 Sumatriptan Iontophoretic Transdermal Patch
- Period 2 (Experimental): NP101 Patch
  Interventions: Drug: NP101 Sumatriptan Iontophoretic Transdermal Patch
- Period 3 (Experimental): NP101 Patch
  Interventions: Drug: NP101 Sumatriptan Iontophoretic Transdermal Patch
- Period 4 (Experimental): NP101 Patch
  Interventions: Drug: NP101 Sumatriptan Iontophoretic Transdermal Patch
- Period 5 (Experimental): NP101 Patch
  Interventions: Drug: NP101 Sumatriptan Iontophoretic Transdermal Patch

INTERVENTIONS:
Drug: NP101 Sumatriptan Iontophoretic Transdermal Patch — NP101 transdermal patch delivering sumatriptan for 4 hours.

SUMMARY:
The primary objective is to compare the pharmacokinetics (PK) profiles among five NP101 patches in healthy volunteers.

The secondary objective is to evaluate the safety of NP101 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian men or women aged 18 to 45.
* Subjects have BMI of 18 to 30 kg/m2 inclusive.
* Subject judged to be in good health, based upon the results of a medical history, physical examination, vital signs, ECG and laboratory profile. Subjects will not have any clinically significant abnormal findings in order to qualify for enrollment.
* Subject must have a negative drug screen at screening and on Day -1 for all treatment.
* Subjects must be nonsmokers, defined as having not used any tobacco products in the 6 months before screening.
* The subjects will have received no other medication except birth control, for two weeks prior to study entry.
* Subjects must have not consumed alcoholic beverages, poppy seeds, grapefruit, and/or grapefruit juice within 72 hours prior to admission.
* Female of childbearing potential must have a negative pregnancy test at screening and on Day -1 for all treatment.
* In the investigator's opinion, the subject must be likely to complete the study.
* Subjects must be able to communicate effectively and be capable of reading and understanding English and voluntarily sign an IRB approved IC agreement.

Exclusion Criteria:

* Subject has a history of allergy or hypersensitivity to any component of the study patch used in this study.
* Subject has any generalized skin irritation or disease including eczema, psoriasis, melanoma, contact dermatitis or acne.
* Subject has a tattoo that might interfere with skin irritation examination.
* Subject has a history of epilepsy or conditions associated with a lowered seizure threshold.
* Subject has a history of basilar or hemiplegic migraines.
* Subject has suspected or confirmed cardiovascular disease that contraindicates participation.
* Subject has Raynaud's disease.
* Subject has a history (within 1 year) or current evidence of drug or alcohol abuse or dependence.
* Subject with a history of malignancy within the past 5 years.
* Subject has clinically significant abnormal laboratory parameters, vital signs or ECG parameters.
* Subject has SGOT/AST, SGPT/ALT, alkaline phosphatase or total bilirubin ≥ 1.5 times the upper limit of normal.
* Subject with a hemoglobin (Hgb) level of less than 7.5 mmol/L.
* Subject is hepatitis B, hepatitis C or HIV positive.
* Subject has taken an MAO inhibitor, preparations containing St. John's Wort, SSRI, SNRI, TCA, triptan or ergot medication, within one month prior to screening.
* Subject is unwilling to discontinue the use of phosphodiesterase type 5 inhibitor, from screening through the End of Study.
* Subject who has been administered an injectable drug, except for local anesthetic or birth control, within 30 days prior to the initial study drug administration.
* Donation of blood or blood products within 8 weeks prior to study entry.
* Receipt of an investigational drug or participation in any clinical study within 90 days prior to study.
* Subject who requires any medication on a regular basis, with the exception of steroidal contraceptives.
* Concurrent use of Rx or OTC medications or natural medicine (herbal) products, with the exception of steroidal contraceptives.
* Female subject who is pregnant, planning a pregnancy during the study, breast feeding; or if of childbearing potential, not using or unwilling to use an effective form of contraception during the study and for a period of 30 days following dosing.
* Subject who is considered to be an unsuitable candidate for receiving sumatriptan, or as being unsuitable for any other reason.
* Subject is electrically sensitive (e.g., prior iontophoresis with adverse outcome related to the current delivered by the device) or who have an implantable electronic device (e.g., pacemaker).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The primary objective was to compare the pharmacokinetics (PK) profiles among five NP101 patches in healthy volunteers. | Blood samples were collected at time points: pre-dose (within 15 minutes prior to dosing) and at 0.25, 0.50, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hrs post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Canas, MD, Principal Investigator — Prism Research
Locations (1):
- Prism Research, Saint Paul, Minnesota, United States